CLINICAL TRIAL: NCT01620294
Title: Abdomen Closure Using Triclosan Coated Absorbable Suture vs Uncoated Sutures of the Same Base Material
Brief Title: Abdominal Wall Closure With Triclosan-coated Suture
Acronym: TCS09
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Medical Center, University of Pecs, Prof. O P Horvath MD, PhD.ScD
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: triclosan-coated-suture2009
Record Dates: First submitted 2010-05-10; First posted 2012-06-15 (Estimated); Last update posted 2012-06-15 (Estimated); Status verified 2012-06

CONDITIONS: Infection
Keywords: surgical site infection; elective colorectal surgery; level of surgical site infection; complication of surgical site infection; type of changed bandage; frequency of bandage changing
MeSH Terms: conditions — Infections; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- triclosan (Experimental): Two arms are separated by computer randomization at abdominal wall closure: application of triclosan-coated and non-coated PDS suture (PDS vs. PDS-Plus).
  Interventions: Procedure: abdominal wall closure
- uncoated (Experimental): Two arms are separated by computer randomization at abdominal wall closure: application of triclosan-coated and non-coated PDS suture (PDS vs. PDS-Plus).
  Interventions: Procedure: surgical site infection

INTERVENTIONS:
Procedure: abdominal wall closure — triclosan-coated (PDS-Plus) and non-coated (PDS) suture to close the abd. wall
  Other Names: presence of surgical site infection; level of surgical site infection
  Arms: triclosan
Procedure: surgical site infection — triclosan-coated (PDS-Plus) and non-coated (PDS) suture to close the abd. wall
  Other Names: presence of surgical site infection; level of surgical site infection
  Arms: uncoated

SUMMARY:
After open colorectal surgery the surgical site infection (SSI) is very high among abdominal surgeries. The goal of the investigators randomized, prospective, multicentric, internet-based study is to compare rate of SSI after surgery of colon and rectum by using triclosan-coated suture for abdominal wall closure. 180-180 cases in seven centres are involved in this study. Two arms are separated by computer randomization at abdominal wall closure: application of triclosan-coated and non-coated PDS suture (PDS versus PDS-Plus). Triclosan is an antiseptic material which the investigators hope will provide better local infection control at the site with reducing the risk of bacterial colonisation.

DETAILED DESCRIPTION:
After open colorectal surgery the surgical site infection (SSI) is very high among abdominal surgeries. The goal of our randomized, prospective, multicentric, internet-based study is to compare rate of SSI after surgery of colon and rectum by using triclosan-coated suture for abdominal wall closure. Two arms are separated by computer randomization at abdominal wall closure: application of triclosan-coated and non-coated PDS suture (PDS versus PDS-Plus). Triclosan is an antiseptic material which we hope provides better local infection control at the site with reducing the risk of bacterial colonisation.

attached website: www.itplan.hu/sebstudy/ Randomizing patients: 1. logging in (completing the ID panel) 2. on-line randomization 3. patient appears on list 4. operation (recording details) 5. recording - post-operation events

* complications
* control examination

ELIGIBILITY:
Inclusion Criteria:

* Elective (subjected to bowel preparation) operations
* Benign or malignant colon or rectal disease
* Age: 18-80
* Bowel opening is made during operation

Exclusion Criteria:

1. Cannot be randomized:

   * Systemic diseases influencing local surgical site healing
   * Insulin-dependent diabetes mellitus
   * Child B-C liver cirrhosis
   * Kidney disease requiring dialysis
   * Immune-suppression treatment
   * IBD
   * Acute surgery or unprepared bowel
   * After being informed patient does not sign the statement of consent
2. To be excluded later:

   * Surgically incurable tumour
   * Septic state or complication occurred in the post-operational stage
   * Patient withdraws the signed consent before the examination is closed
3. Undesirable complication:

   * Sterile surgical site separation
   * Suture break during the post-operational stage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
quality and quantity of wound discharge | 30 days

SECONDARY OUTCOMES:
number of applied different types of bandages | 30 days
charges of wound care | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Ors Peter Horvath, MD, PhD, DSc, Principal Investigator — Head of Surg.Dept. Univ. of Pecs, Hungary - ophorvath@iseb.pote.hu
Locations (1):
- Department of Surgery Medical Faculty, University of Pecs, Hungary, Pécs, Hungary

REFERENCES:
- [Background] Mangram AJ, Horan TC, Pearson ML, Silver LC, Jarvis WR. Guideline for prevention of surgical site infection, 1999. Hospital Infection Control Practices Advisory Committee. Infect Control Hosp Epidemiol. 1999 Apr;20(4):250-78; quiz 279-80. doi: 10.1086/501620. No abstract available. PMID 10219875
- [Background] Nishikawa K, Hanyuu N, Yuda M, Tanaka Y, Matsumoto A, Yasue H, Hayashi T, Kawano S, Usuba T, Iino T, Mizuno R, Iwabuchi S. How can we control intraoperative bacterial contamination and surgical-site infection during an anterior resection or Hartmann's/Miles' operation? J Gastrointest Surg. 2008 Nov;12(11):1995-2000. doi: 10.1007/s11605-008-0582-z. Epub 2008 Jul 18. PMID 18636300
- [Background] Watanabe A, Kohnoe S, Shimabukuro R, Yamanaka T, Iso Y, Baba H, Higashi H, Orita H, Emi Y, Takahashi I, Korenaga D, Maehara Y. Risk factors associated with surgical site infection in upper and lower gastrointestinal surgery. Surg Today. 2008;38(5):404-12. doi: 10.1007/s00595-007-3637-y. Epub 2008 Apr 30. PMID 18560962
- [Background] Kobayashi M, Mohri Y, Inoue Y, Okita Y, Miki C, Kusunoki M. Continuous follow-up of surgical site infections for 30 days after colorectal surgery. World J Surg. 2008 Jun;32(6):1142-6. doi: 10.1007/s00268-008-9536-6. PMID 18338205
- [Background] Nichols RL, Choe EU, Weldon CB. Mechanical and antibacterial bowel preparation in colon and rectal surgery. Chemotherapy. 2005;51 Suppl 1:115-21. doi: 10.1159/000081998. PMID 15855756
- [Background] Barbolt TA. Chemistry and safety of triclosan, and its use as an antimicrobial coating on Coated VICRYL* Plus Antibacterial Suture (coated polyglactin 910 suture with triclosan). Surg Infect (Larchmt). 2002;3 Suppl 1:S45-53. doi: 10.1089/sur.2002.3.s1-45. PMID 12573039
- [Background] Fleck T, Moidl R, Blacky A, Fleck M, Wolner E, Grabenwoger M, Wisser W. Triclosan-coated sutures for the reduction of sternal wound infections: economic considerations. Ann Thorac Surg. 2007 Jul;84(1):232-6. doi: 10.1016/j.athoracsur.2007.03.045. PMID 17588420
- [Background] Justinger C, Moussavian MR, Schlueter C, Kopp B, Kollmar O, Schilling MK. Antibacterial [corrected] coating of abdominal closure sutures and wound infection. Surgery. 2009 Mar;145(3):330-4. doi: 10.1016/j.surg.2008.11.007. Epub 2009 Jan 25. PMID 19231586